CLINICAL TRIAL: NCT00670098
Title: Psychosocial Changes Associated With Weight Loss
Brief Title: Changes in Sexual Function Following Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: DK72452; R01DK072452 (NIH)
Record Dates: First submitted 2008-04-30; First posted 2008-05-01 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2011-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: Bariatric surgery
- 2 (Experimental)
  Interventions: Behavioral: lifestyle intervention (behavioral weight loss)

INTERVENTIONS:
Procedure: Bariatric surgery — patients receive either gastric bypass or lap-band
  Arms: 1
Behavioral: lifestyle intervention (behavioral weight loss) — participants attend biweekly weight loss counseling group sessions
  Arms: 2

SUMMARY:
The main purposes of the study are to compare changes in sexual function, changes in sex hormones, and changes in body image and marital satisfaction at 12, 24, 36 and 48 months postoperatively in two groups: individuals who undergo a bariatric surgical procedure and extremely obese individuals with similar obesity-related comorbidities who do not seek surgery (treatment comparison group).

The mechanisms by which extreme obesity affects sexual functioning have received little attention. Recent epidemiologic studies suggest that obesity and physical inactivity are independently related to the likelihood of developing sexual dysfunction over time. For example, men with a BMI greater than 29 kg/m2 have a 30% greater risk of developing erectile dysfunction and up to 50 % of ED cases can be attributed to hypertension and cardiovascular disease, both commonly associated with obesity. Many treatments for hypertension have also been shown to interfere with sexual function.

Changes in sex hormones with increasing BMI have not received much attention either. Obesity has been associated with decreases in testosterone and sex hormone binding globulin for men and increases in testosterone and estrogen for women. Several studies have shown improvement in sex hormone levels in both men and women following weight loss. Sexual functioning has never been assessed in association with weight loss and whether through improvements in body image, sex hormones, or obesity related comorbidities, bariatric surgery may have a profound effect on sexual functioning.

Dr. Ray Rosen, the Principal investigator for this sub study, has conducted a previous investigation focused on sexual functioning after weight loss in a behavioral weight loss program. Specifically, he looked at short and long term sexual function outcomes associated with Type-2 diabetes. His previous work in this area has shown that patients are willing to participate in studies of sexual function.

The Psychosocial Changes study assesses sexual function in two ways. Participants first fill out a packet of questionnaires covering topics related to depression, quality of life, body image, and marital and sexual functioning. They also give a blood sample in order for us to assess levels of sex hormones including testosterone, luteinizing hormone, estradiol, follicle stimulating hormone, and others.

ELIGIBILITY:
Inclusion Criteria:

* • Age: Patients must be between 18 and 65 years of age.

  * Gender: Both women and men are eligible to participate.
  * Ethnicity and Race: Individuals from all ethnic and racial groups will be invited to participate.
  * Body Mass Index: 40 to 60 kg/m2 (or of > 35 kg/m2 in the presence of co-morbid medical conditions).
  * Ambulation: Patients must be ambulatory, given the frequent number of assessments (and difficult arranging transportation for non-ambulatory individuals
  * Competent: The patient must be able to communicate with the investigator and be legally competent, provide written informed consent.

Exclusion Criteria:

* • Any major illnesses that the surgical team believes present too great a risk for surgery. These include severe cardiac and pulmonary diseases, as well as uncontrolled type 2 diabetes.

  * Evidence of major depression or other psychiatric disorder (schizophrenia, bipolar disorder, major depression, bulimia nervosa, etc.) that significantly interferes with daily living and functioning.
  * Use of medications known to significantly increase body weight, such as systemic steroids or psychiatric medications including lithium, tricyclic antidepressants, and anti-psychotic agents (The use of selective serotonin re-uptake inhibitors (SSRIs) will not be excluded because of their widespread use and lesser effect on body weight.)
  * Patients who are not in an ongoing romantic relationship
  * Any current (past 12 months) substance abuse or dependence disorder.
  * Pregnancy or lactation (Those who are pregnant do not undergo bariatric surgery. In addition, the hormone changes induced by pregnancy are known to interfere with the hormones examined in this study, confounding the findings. Participants who become pregnant while in this study will be withdrawn from the study.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2005-08; Primary Completion 2007-10 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Sexual functioning as measured by the International Index for Erectile Dysfunction (for men) and the Female Sexual Function Inventory (for women) | 48 months

SECONDARY OUTCOMES:
sex hormones | 48 months
body image (Body Shape Questionnaire and The Body Image Quality of Life Questionnaire) | 48 months
relationship functioning (Dyadic Adjustment Scale) | 48 months
quality of life (Impact of Weight on Quality of Life questionnaire and Medical Short Form Survey) | 48 months

REFERENCES:
- [Derived] Sarwer DB, Spitzer JC, Wadden TA, Mitchell JE, Lancaster K, Courcoulas A, Gourash W, Rosen RC, Christian NJ. Changes in sexual functioning and sex hormone levels in women following bariatric surgery. JAMA Surg. 2014 Jan;149(1):26-33. doi: 10.1001/jamasurg.2013.5022. PMID 24190440